CLINICAL TRIAL: NCT06645977
Title: Prospective Observational Study of Patients With Interstitial Lung Disease (RESPIRARE)
Brief Title: Patients With Interstitial Lung Disease
Acronym: RESPIRARE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6393
Record Dates: First submitted 2024-03-18; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective monocentric collection of data from adult patients with interstitial lung disease (ILD), to provide real-world data on current patient management at the ILD clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of ILD, according to international guidelines.

Exclusion Criteria:

* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with interstitial lung disease from ILD clinic of the Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-04 (Estimated); Study Completion 2025-04-04 (Estimated)

PRIMARY OUTCOMES:
Prevalce ILD | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, RM, Italy